CLINICAL TRIAL: NCT06422858
Title: Sequential Tegafur-gimeracil-oteracil Potassium Capsule (s-1) and Serplulimab Following Concurrent Chemoradiotherapy in the Treatment of Locally Advanced Inoperable Esophageal Squamous Cell Carcinoma: A Single-Arm Phase II Clinical Trial
Brief Title: Sequential Tegafur-gimeracil-oteracil Potassium Capsule (s-1) and Serplulimab Following Concurrent Chemoradiotherapy for Esophageal Squamous Cell Carcinoma
Acronym: Stars
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Principal Investigator, Ji Yongling, PI, Zhejiang Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: STARS-CCRT-ESCC
Record Dates: First submitted 2024-05-09; First posted 2024-05-21 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2024-05

CONDITIONS: Locally Advanced Inoperable Esophageal Squamous Cell Carcinoma
MeSH Terms: interventions — Radiotherapy; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Serplulimab and S1 Chemotherapy Post-Concurrent Chemoradiation (Experimental)
  Interventions: Drug: Serplulimab; Drug: Tegafur-gimeracil-oteracil potassium capsule(S1); Radiation: Radiotherapy; Drug: Cisplatin

INTERVENTIONS:
Drug: Serplulimab — Serplulimab will be administered as a fixed dose of 300 mg via intravenous infusion every three weeks, continuing for up to 12 months or until disease progression, unacceptable toxicity, or withdrawal of consent
Drug: Tegafur-gimeracil-oteracil potassium capsule(S1) — S1 will be administered at a dose of 60 mg/m2 per day, taken orally in two divided doses on day 1 concurrent with radiotherapy, repeated every 28 days; and from day 1 to day 14 of each 21-day cycle, for up to 12 months or until disease progression, unacceptable toxicity, or withdrawal of consent
Radiation: Radiotherapy — Radiotherapy will be delivered as a total dose of 50.4 Gy in 28 fractions over six weeks using techniques such as IGRT, IMRT, VMAT, or TOMO, targeting the primary tumor and associated lymph nodes
Drug: Cisplatin — Cisplatin will be administered at a dose of 75 mg/m^2 on day 1 concurrent with radiotherapy, repeated every 28 days

SUMMARY:
This Phase II trial evaluates the efficacy and safety of Serplulimab combined with S1 chemotherapy in patients with inoperable, locally advanced esophageal squamous cell carcinoma after concurrent chemoradiation. The primary endpoint is the one-year progression-free survival rate. Secondary measures include clinical response rates, overall survival, duration of response, and safety profiles. Exploratory goals focus on the potential of biomarkers like PD-L1 and ctDNA to predict treatment outcomes. Treatment involves initial chemoradiation followed by consolidation with Serplulimab and S1, continuing for up to 12 months or until disease progression or unacceptable toxicity.

DETAILED DESCRIPTION:
Detailed Description:

This single-arm, Phase II study is designed to assess the efficacy and safety of the combination of Serplulimab (an anti-PD-1 antibody) and S1 (an oral fluoropyrimidine derivative) in patients with locally advanced, inoperable esophageal squamous cell carcinoma (ESCC), following concurrent chemoradiation therapy.

Study Treatment Regimen:

Patients enrolled in the study will first undergo concurrent chemoradiation, which includes a total radiation dose of 50.4 Gy delivered in 28 fractions over six weeks. Radiation will be administered using modern techniques such as image-guided radiation therapy (IGRT), intensity-modulated radiation therapy (IMRT), volumetric modulated arc therapy (VMAT), or helical tomotherapy (TOMO), ensuring precise targeting of the tumor and surrounding lymph nodes. Concurrent chemotherapy consists of cisplatin (75 mg/m2 on day 1) and S1 (60 mg/m2 per day, given in two divided doses from day 1 to day 14, repeated every 28 days).

Following chemoradiation, patients will receive consolidation therapy with Serplulimab administered at a fixed dose of 300 mg every three weeks via intravenous infusion, alongside S1 (60 mg/m2 per day, on days 1-14 of a 21-day cycle). This consolidation phase will continue for up to 12 months or 17 cycles, unless there is disease progression, patient withdrawal, onset of unacceptable toxicity, or initiation of new anti-cancer treatment.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand and voluntarily sign a written informed consent form, which must be signed before initiating any study-specific procedures.
* Male or female participants aged between 18 and 70 years at the time of informed consent.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1. Histologically or cytologically confirmed diagnosis of locally advanced esophageal squamous cell carcinoma (ESCC); or patients who refuse surgery; staged as T1-4bN1-3M0 (according to AJCC 8th edition).
* Medically inoperable or refusal of surgery.
* No prior anti-tumor treatment.
* Expected survival of at least 6 months.
* At least one measurable lesion as defined by RECIST v1.1.
* Participants must provide either archived (within the last 2 years) or freshly obtained tumor tissue samples, with at least three unstained FFPE pathology slides.
* Adequate organ function defined as follows:

  a. Hematology (no blood transfusions or growth factor support within 7 days before starting study treatment): i. Absolute Neutrophil Count (ANC) ≥1.5×10^9/L (1500/mm³); ii. Platelet count ≥100×10^9/L (100000/mm³); iii. Hemoglobin ≥90 g/L. b. Renal: i. Calculated creatinine clearance (CrCl) ≥50 mL/min using the Cockcroft-Gault formula: CrCl (mL/min) = {(140-age) × weight (kg) × F} / (SCr (mg/dL) × 72), where F=1 for males and 0.85 for females; SCr=serum creatinine.

ii. Urinary protein <2+ or 24-hour urinary protein quantification <1.0 g. c. Liver: i. Total bilirubin (TBiL) ≤1.5×ULN; ii. AST and ALT ≤2.5×ULN (≤5×ULN for participants with liver metastases); iii. Serum albumin (ALB) ≥28 g/L. d. Coagulation: International Normalized Ratio (INR) and Activated Partial Thromboplastin Time (APTT) ≤1.5×ULN, unless the participant is receiving anticoagulant therapy and INR and APTT are within the expected range of their therapeutic use.

e. Cardiac: Left Ventricular Ejection Fraction (LVEF) ≥50%.

* Female participants of childbearing potential must have a negative urine or serum pregnancy test within 3 days prior to the first dose of study medication. If urine test is not conclusive, a serum test will be administered. If sexually active with a non-sterilized male partner, the participant must agree to use effective contraception during the study and for 120 days after the last dose of study medication. Discussion with the researcher is required regarding cessation of contraception after this point.
* Male participants with female partners of childbearing potential must agree to use effective contraception from screening to 120 days after the last dose of study medication. Discussion with the researcher is required regarding cessation of contraception after this point.
* Willing and able to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures.

Exclusion Criteria:

* Previous anti-tumor treatment (including chemotherapy, radiation therapy, surgery, or immunotherapy).
* Initial diagnosis with metastases to vital organs such as the liver, bones, lungs, brain, adrenal glands, etc. (stage IVb esophageal cancer).
* History of thoracic radiotherapy.
* Presence of an esophageal mediastinal fistula and/or esophageal tracheal fistula before treatment.
* Known or suspected allergy to any component of S1, serplulimab, or cisplatin.
* Pregnant or breastfeeding women.
* Inability to provide informed consent due to psychological, familial, or social reasons.
* History of any malignancy other than esophageal cancer within the past 5 years, except for adequately treated non-melanoma skin cancer, in-situ cervical cancer, or cured early-stage prostate cancer.
* Unable to tolerate chemoradiation due to severe cardiac, pulmonary, hepatic, renal dysfunctions, hematological diseases, or cachexia.
* Active autoimmune diseases, history of autoimmune diseases (including but not limited to colitis, hepatitis, hyperthyroidism, or syndromes), history of immunodeficiency (including positive HIV test), or other acquired or congenital immunodeficiency diseases, history of organ transplant or allogeneic bone marrow transplant.
* Active hepatitis B (HBV DNA ≥ 2000IU/mL or 10×10^4 copies/mL), positive hepatitis C antibody with elevated HCV RNA levels above the lower limit of detection.

History of immunodeficiency; positive HIV antibody; current long-term use of systemic corticosteroids or other immunosuppressants.

* Serious infection within 4 weeks before the first administration of study medication, including but not limited to complications requiring hospitalization, sepsis, or severe pneumonia; active infection requiring systemic anti-infective treatment within 2 weeks before the first dose (excluding antiviral treatment for hepatitis B or C).

Known active tuberculosis (TB), suspected active TB requiring clinical exclusion; known active syphilis infection.

* Vaccination with live or attenuated live vaccines within 30 days before the first dose of study medication or planning to receive such vaccines during the study period; inactivated vaccines are permitted.
* History of interstitial lung disease or non-infectious pneumonia.
* History of myocarditis, cardiomyopathy, malignant arrhythmias, unstable angina, myocardial infarction within the past 12 months, congestive heart failure as determined by NYHA Class II or higher, or vascular diseases such as aortic aneurysm at risk of rupture, or other cardiac damage that could compromise the safety evaluation of the study medication (such as poorly controlled arrhythmia or myocardial ischemia).
* Known history of mental illness, drug abuse, alcoholism, or drug addiction.
* Non-malignant systemic diseases or symptoms secondary to tumors that could pose a higher medical risk or confound the assessment of survival, such as leukemic reaction (white cell count >20×10^9/L) or cachexia manifestations (known weight loss exceeding 10% in the 3 months prior to screening).
* Any condition that, in the opinion of the investigator, might pose a risk to the participant, interfere with the evaluation of the study medication, or confound the interpretation of study results.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2024-05-20 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
One-Year Progression-Free Survival (PFS) | 1 year
  The primary outcome measure is the proportion of participants who are alive and free from disease progression at one year after initiating treatment. Progression is defined according to RECIST v1.1 criteria as a 20% increase in the sum of diameters of target lesions, the appearance of new lesions, or the worsening of non-target disease

SECONDARY OUTCOMES:
Incidence of Clinical Complete Response Rate (cCR) at 3 months after treatment initiation | Assessed at 3 months after treatment initiation
  The rate of participants achieving a clinical complete response assessed by RECIST v1.1 criteria. A clinical complete response is defined as the disappearance of all target lesions and normalization of tumor marker levels.
Overall Survival (OS) | From the start of treatment up to 3 years
  Overall survival is defined as the time from the start of treatment to the date of death from any cause. If a patient is not known to have died, survival time will be censored at the date of the last known follow-up.
Duration of Response (DoR) | From the first documented response up to 2 years
  Duration of response is measured from the time measurement criteria are first met for Complete Response or Partial Response (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented.
Incidence of Treatment-Emergent Adverse Events | Throughout the study, estimated at 12 months
  The incidence and severity of adverse events categorized by the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 5.0.
EORTC-QoL-C30 Score(Quality of Life) | At baseline, 6 months, and 12 months
  Qualitasured using validated instruments such as the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC-QLQ-C30). The quality of life score is calculated based on the rules set by EORTC (range 0-100). A lower score indicates better quality of life on the symptom scales, while a higher score indicates better quality of life scores on the overall health and functional scales.

OTHER OUTCOMES:
Grade 3 Pneumonia Incidence [Safety and Tolerability] | through study completion, an average of 1 year
  The study will implement a pre-specified safety threshold where if the incidence of Grade 3 pneumonia, as categorized by the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), exceeds 15% of participants, the trial may be modified or halted to assess and mitigate risks to patient safety.

CONTACTS AND LOCATIONS:
Overall Officials: Yongling Ji, Principal Investigator — Zhejiang Cancer Hospital
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No